CLINICAL TRIAL: NCT00005246
Title: Epidemiology of Insulin and Dehydroepiandrosterone Sulfate and Coronary Heart Disease Mortality
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1128; R01HL041785 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To determine whether serum insulin is a risk factor for coronary heart disease morbidity and mortality and whether dehydroepiandrosterone sulfate (DHEAS) is a risk factor for coronary heart disease mortality. Also, to ascertain the determinants of serum insulin levels among middle-aged men.

DETAILED DESCRIPTION:
BACKGROUND:

In 1972, the Multiple Risk Factor Intervention Trial began recruiting 12,866 men, ages 35 to 57, selected for elevation of one or more risk factors but free from coronary heart disease and followed them for an average of seven years after randomization to a risk factor modification group or to a control group referred to their own physicians for treatment. The serum from MRFIT had been stored since 1972. Detailed follow-up for the cohort was completed through 1985 and was extended through 1988 using the National Death Index.

The role of insulin as a major risk factor for atherosclerosis resurfaced in the 1980s and was the subject of much research at the basic science, clinical, and epidemiological levels. The MRFIT serum data base probably was the only remaining such serum bank in the United States that could test the relationship between insulin levels and coronary heart disease mortality that included detailed measurements of other major cardiovascular risk factors, as well as both baseline and two-hour post-load glucose levels in a predominantly non-diabetic population.

DHEAS is the most abundant circulating steroid hormone in man and is readily converted to DHEA which is a potent non-competitive inhibitor of glucose-6-phosphate dehydrogenase, the rate limiting enzyme of the pentose cycle. Several studies suggest a key role of DHEAS in obesity, lipid metabolism, cellular proliferation, and atherosclerosis. Barrett-Connor in 1986 reported that low levels of this hormone were a risk factor for cardiovascular disease in men. Other studies report that administration of DHEAS to laboratory animals appears to delay aging, prevent obesity, and lower serum cholesterol levels.

DESIGN NARRATIVE:

A nested case-control study was conducted using the stored blood serum. Laboratory measurements were done blindly without knowledge of whether the specimen was from a case or a control. Insulin was measured in all 600 specimens. DHEAS was measured in 200 cases and 100 controls. The means and distribution of insulin or DHEAS levels were compared between cases and controls. The analysis was done separately for the coronary heart disease deaths and surviving myocardial infarction cases and, if there were no differences between the case groups, they were pooled for comparison with the controls. The relationships were determined among the potential confounders, coronary heart disease morbidity and mortality and serum insulin or DHEAS levels. This analysis also included data on baseline serum cholesterol, systolic and diastolic blood pressure, cigarette smoking, serum thiocyanate, HDL and LDL cholesterol, triglycerides, basal metabolic index, fasting and one-hour blood glucose. Alcohol intake, physical activity, pulmonary function, and education were also evaluated. The relationships among insulin or DHEAS and coronary heart disease morbidity and mortality were evaluated after adjusting for possible confounders.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-08; Study Completion 1991-07 (Actual)

REFERENCES:
- [Background] Kuller LH, Eichner JE, Orchard TJ, Grandits GA, McCallum L, Tracy RP. The relation between serum albumin levels and risk of coronary heart disease in the Multiple Risk Factor Intervention Trial. Am J Epidemiol. 1991 Dec 1;134(11):1266-77. doi: 10.1093/oxfordjournals.aje.a116030. PMID 1755441
- [Background] Eichner JE, Kuller LH, Orchard TJ, Grandits GA, McCallum LM, Ferrell RE, Neaton JD. Relation of apolipoprotein E phenotype to myocardial infarction and mortality from coronary artery disease. Am J Cardiol. 1993 Jan 15;71(2):160-5. doi: 10.1016/0002-9149(93)90732-r. PMID 8421977